CLINICAL TRIAL: NCT05257252
Title: The Effect of "Persons With Disability Friendly Nursing Education Program" on Nursing Students' Emphatic Tendency and Perception of Caring Competency
Brief Title: The Effect of "Persons With Disability Friendly Nursing Education Program"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Prof. Dr., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/386
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Nurse-Patient Relations; Nurse's Role; Nursing Caries
Keywords: Disability; Nursing education; Persons with disability

STUDY DESIGN:
Intervention Model Description: Randomized controlled pretest- post test experimental design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Persons With Disability Friendly Nursing Education Program" (Experimental): Intervention group after determining the students according to the research criteria, they were randomized into intervention and control groups. Firstly, pre-tests were applied to the students in the experimental group.
  Interventions: Behavioral: "Persons With Disability Friendly Nursing Education Program"
- non-"Persons With Disability Friendly Nursing Education Program" (No Intervention): Firstly, Pre-tests were applied to the students in the control group. No intervention was applied to this group. Posttests were made 3 months after pre-test.

INTERVENTIONS:
Behavioral: "Persons With Disability Friendly Nursing Education Program" — Persons With Disability Friendly Nursing Education Program developed based on the Story Theory, 2 weeks program
  Arms: "Persons With Disability Friendly Nursing Education Program"

SUMMARY:
The purpose of this research; The aim of this study is to measure the effect of the Persons With Disability Friendly Nursing Education Program developed based on the Story Theory on the empathic tendencies of senior nursing students towards persons with disability and their perceptions of competence of senior nursing students to care for persons with disability. In the research, a multi-stage evaluation design from mixed method research will be used. Focus group interviews will be conducted before and after the program in the qualitative dimension of the research, while the randomized controlled double-blind pretest-posttest control group experimental design will be used in the quantitative dimension. The data of the research will be collected in the Department of Nursing of the Faculty of Health Sciences of Ondokuz Mayis University in Samsun, Turkey.

DETAILED DESCRIPTION:
The purpose of this research; The aim of this study is to measure the effect of the Persons With Disability Friendly Nursing Education Program developed based on the Story Theory on the empathic tendencies of senior nursing students towards persons with disability and their perceptions of competence of senior nursing students to care for persons with disability. In the research, a multi-stage evaluation design from mixed method research will be used. Focus group interviews will be conducted before and after the program in the qualitative dimension of the research, while the randomized controlled double-blind pretest-posttest control group experimental design will be used in the quantitative dimension. The data of the research will be collected in the Department of Nursing of the Faculty of Health Sciences of Ondokuz Mayis University in Samsun, Turkey. The program will be applied to nursing senior students in this department. Before the training program, focus group discussions will be held with nursing students, and the content of the training program will be created. The pre-test data of the study will be collected using an introductory information form questioning sociodemographic characteristics, Efficacy Perceptions Form for Caring for Persons with Disabilities, Empathic Tendency Scale and Achievement Test. A 2-week " Persons With Disability Friendly Nursing Education Program" will be applied to the experimental group. After the program, focus group discussions will be held with the students in the experimental group, and the program will be evaluated. Post-tests will be applied to the experimental and control groups 3 months after the program. Descriptive statistics, paired t-test, chi-square, Mann-Whitney U, Wilcoxon analysis will be used in the analysis of the data. Content analysis will be used in qualitative data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being senior nursing student

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Empathic Tendency Scale | 3 month
  The Empathic Tendency Scale was developed by Dokmen (1988). The scale consists of 20 items, which are answered with a five-point rating (1= totally contradictory, 5= totally appropriate). 12 items of the scale consist of positive statements and 8 items of negative statements. Negative statements are reverse coded. The pupae that can be taken from the scale are between 20 and 100 points. High scores mean high empathic tendency. Dokmen (1988) found the reliability coefficient of the scale as .72 in his study.
Form of Perceptions for Caring for Persons with Disabilities | 3 month
  Form of Perceptions for Caring for Persons with Disabilities will be evaluated with a 20-item scale developed by researchers in line with the literature and scored between 0-10 (0, I don't feel adequate at all; 10, I feel very competent). Students will express their perceptions of competence by scoring from 0 to 10 on this scale. Higher scores indicate higher perceptions of caregiving competence.
Program Achievement Test | 3 month
  The Achievement Test is a test consisting of 20 closed-ended questions with 5 answer options, developed by the researchers in line with the information in the training program. The increase in the scores obtained from the achievement test indicates that the perception of efficacy towards caregiving increases. In the test, each correct answer corresponds to "1" point and each wrong answer corresponds to "0" point.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Aydın Avci, Prof. Dr., Study Director — Ondokuz Mayıs University
Locations (1):
- Güven Soner, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No